CLINICAL TRIAL: NCT05029622
Title: A Phase III, Open-label, Multicentre, Single Arm Study to Assess the Efficacy and Safety of the Triptorelin 6-month Formulation in Chinese Paediatric Participants With Central Precocious Puberty.
Brief Title: A Study to Assess the Efficacy and Safety of the Triptorelin 6-month Formulation in Paediatric Participants With Central Precocious Puberty.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-CN-52014-244; 2022-003857-78 (EudraCT Number)
Record Dates: First submitted 2021-08-09; First posted 2021-08-31 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triptorelin formulation for Intramuscular injection (IM). (Experimental)
  Interventions: Drug: Triptorelin Pamoate

INTERVENTIONS:
Drug: Triptorelin Pamoate — Triptorelin 6-month formulation for IM on day 1 and Month 6.

SUMMARY:
The purpose of the protocol is to assess the efficacy of the triptorelin 6 month PR (Prolonged Release) formulation in suppressing LH (Luteinising hormone) levels to prepubertal levels (defined as a peak LH ≤5 IU/L) after i.v. GnRH (Gonadotropin-releasing Hormone) stimulation at Month 6 (Day 169) in Chinese children with CPP (Central Precocious Puberty).

ELIGIBILITY:
Inclusion Criteria:

* Participant is less than 9 years old for girls and less than 10 years old for boys at initiation of triptorelin treatment or at the time of signing the informed consent.
* Participant must present evidence of CPP documented by:
* Onset of development of secondary sex characteristics (breast development in girls or testicular enlargement in boys according to the Tanner method: Stage II) before the age of 8 years in girls and 9 years in boys.
* Pubertal response of LH to GnRH stimulation test (stimulated peak LH ≥6 IU/L) in both sexes.
* Difference between bone age (BA) and CA >1 year.
* Girls with Tanner staging ≥2 for breast development and who have enlarged uterine length and/or ovarian volume and at last 2 follicles with diameter >4 mm in the ovary observed by pelvic type B ultrasound at the Screening visit; boys who have testicular volume ≥4 mL observed by testicular orchidometer at the Screening visit.
* Girls who have already had menophania/menarche must have a negative highly sensitive (urine) pregnancy test as required by local regulations within 24 hours before the first dose of study intervention and should not be at risk of pregnancy throughout the study period.

Exclusion Criteria:

* Gonadotropin-independent (peripheral) precocious puberty: extrapituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroid secretion.
* Non-progressing isolated premature thelarche.
* Presence of an unstable intracranial tumour or an intracranial tumour requiring neurosurgery or cerebral irradiation. Participants with hamartomas not requiring surgery are eligible.
* Prior or current therapy with a GnRHa (Gonadotropin-releasing Hormone Agonist) , medroxyprogesterone acetate, growth hormone or insulin-like growth factor 1 (IGF 1).Use of anticoagulants (heparin and coumarin derivatives) within the 2 weeks prior to the Screening visit.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (14):
- China (14):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - No.1 Hospital of Jilin University (Bethune first hospital of Jilin University), Changchun
  - Children's Hospital of Fudan University, Changhai
  - Hunan children's hospital, Changsha
  - Chengdu Women's & Children's Central Hospital, Chengdu
  - Shandong Provincial Hospital, Jinan
  - Linyi Maternal and Child Health Care Hospital, Linyi
  - Jiangxi Provincial Children's Hospital, Nanchang
  - Pingxiang Maternity and Child Care, Pingxiang
  - Children's Hospital of Soochow University, Suzhou
  - Wuhan Children's Hospital Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan
  - Wuxi children's Hospital, Wuxi
  - Zhengzhou Children's Hospital , Henan Children's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Yu X, Cheng X, Wei H, Xu X, Gong C, Li G, Yao H, Zhou L, Zhong Y, Yang Y, Luo F, Zhang Y, Huang F, Shi X, Cabri P, Luo X. A Phase 3, Open-Label, Single-Arm Trial of the Efficacy and Safety of Triptorelin 6-Month Formulation in Chinese Children with Central Precocious Puberty. Adv Ther. 2024 Dec;41(12):4537-4556. doi: 10.1007/s12325-024-02991-x. Epub 2024 Oct 16. PMID 39412628
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2024/08/08212539/D-CN-52014-244-lay-results-summary-1.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open-label, single arm, study was conducted in children with central precocious puberty (CPP) at 12 investigational sites in China from 25 August 2021 to 13 February 2023.
Pre-assignment Details: This study consisted of screening period (up to 28 days) and study duration of minimum 12 months and up to 13 months including screening period.
Groups:
- All Participants: Participants received triptorelin pamoate 22.5 milligrams (mg) intramuscular (IM) injection on Day 1.
Period: Overall Study
Arm/Group | All Participants
Started | 66
Completed | 65
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population consisted of all participants who received at least 1 dose of study intervention.
Groups:
- All Participants: Participants received triptorelin pamoate 22.5 mg IM injection on Day 1.
Arm/Group | All Participants
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Luteinising Hormone (LH) Suppression
Description: LH response was defined as a peak LH <=5 international units per liter (IU/L) after intravenous (IV) gonadotropin-releasing hormone (GnRH) stimulation. The GnRH stimulation test was performed by using an IV injection of gonadorelin (synthetic GnRH) to stimulate gonadotrophin release and blood samples were collected after the gonadorelin injection for central assessment of serum LH levels. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Month 6
Population: The ITT population consisted of all participants who received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentage of participants | 100 [94.6 to 100.0]

2. Secondary Outcome: Percentage of Participants With LH Response to GnRH Test
Description: LH response was defined as a peak LH <=5 IU/L after IV GnRH stimulation. The GnRH stimulation test was performed by using an IV injection of gonadorelin (synthetic GnRH) to stimulate gonadotrophin release and blood samples were collected after the gonadorelin injection for central assessment of serum LH levels. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Months 3 and 12
Population: The ITT population consisted of all participants who received at least 1 dose of study intervention. Only data from the participants analyzed were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentage of participants
  Month 3: number analyzed (Participants) | 64
  Month 3 | 97.0 [89.5 to 99.6]
  Month 12: number analyzed (Participants) | 65
  Month 12 | 98.5 [91.8 to 100.0]

3. Secondary Outcome: Change From Baseline in Basal Serum LH and Follicle-Stimulating Hormone (FSH) Levels
Description: Basal LH and FSH serum concentrations were analyzed centrally. Change from baseline was defined as the values for LH and FSH at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline and at Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | All Participants
Number analyzed (Participants) | 66
IU/L
  LH, Month 3: number analyzed (Participants) | 64
  LH, Month 3 | -1.6420 (2.4287)
  LH, Month 6 | -1.8015 (2.4109)
  LH, Month 9: number analyzed (Participants) | 57
  LH, Month 9 | -1.6307 (2.3396)
  LH, Month 12: number analyzed (Participants) | 65
  LH, Month 12 | -1.8504 (2.4524)
  FSH, Month 3: number analyzed (Participants) | 64
  FSH, Month 3 | -2.9938 (1.9450)
  FSH, Month 6 | -2.4871 (2.0414)
  FSH, Month 9: number analyzed (Participants) | 57
  FSH, Month 9 | -2.8586 (1.9310)
  FSH, Month 12: number analyzed (Participants) | 65
  FSH, Month 12 | -2.5348 (1.9162)

4. Secondary Outcome: Change From Baseline in Peak Serum LH and FSH Level After the GnRH Stimulation Test
Description: Peak LH and FSH serum concentrations were analyzed centrally. Change from baseline was defined as the values for LH and FSH at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered. Blood samples were collected prior to gonadorelin injection (timepoint T0) and at 30 minutes (T30), 60 minutes (T60) and 90 minutes (T90) after a single IV injection of gonadorelin. A suppressed LH response to GnRH stimulation test was defined as peak serum LH <=5 IU/L among the four timepoints (T0, T30, T60 and T90). The FSH response to GnRH stimulation was the peak serum FSH level among the four timepoints (T0, T30, T60 and T90).
Time Frame: Baseline and at Months 3, 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | All Participants
Number analyzed (Participants) | 66
IU/L
  LH, Month 3: number analyzed (Participants) | 64
  LH, Month 3 | -26.0075 (19.8863)
  LH, Month 6 | -26.2867 (20.3004)
  LH, Month 12: number analyzed (Participants) | 65
  LH, Month 12 | -26.6065 (20.5680)
  FSH, Month 3: number analyzed (Participants) | 64
  FSH, Month 3 | -11.7297 (5.1787)
  FSH, Month 6 | -10.0656 (5.0160)
  FSH, Month 12: number analyzed (Participants) | 65
  FSH, Month 12 | -10.1645 (5.2442)

5. Secondary Outcome: Percentage of Participants With LH Response (Peak LH <=5 IU/L) From Month 6 to Month 12
Description: Peak LH serum concentration was analyzed centrally. LH response was defined as a peak LH <=5 IU/L after IV GnRH stimulation. The GnRH stimulation test was performed by using an IV injection of gonadorelin (synthetic GnRH) to stimulate gonadotrophin release and blood samples were collected after the gonadorelin injection for central assessment of peak LH levels. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: Month 6 to Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 65
percentage of participants | 98.5 [91.8 to 100.0]

6. Secondary Outcome: Percentage of Participants With Prepubertal Levels of Sex Steroids
Description: Prepubertal sex steroids assessment included estradiol in female participants and testosterone in male participants. Prepubertal sex steroids levels were defined as: estradiol <=20 picogram (pg)/ milliliter (mL) in female participants and testosterone <=30 nanogram (ng)/ deciliter (dL) in male participants. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Months 3, 6, 9 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentage of participants
  Month 3: number analyzed (Participants) | 64
  Month 3 | 97.0 [89.5 to 99.6]
  Month 6 | 100 [94.6 to 100.0]
  Month 9: number analyzed (Participants) | 57
  Month 9 | 86.4 [75.7 to 93.6]
  Month 12: number analyzed (Participants) | 65
  Month 12 | 98.5 [91.8 to 100.0]

7. Secondary Outcome: Change From Baseline in Mean Height for Age (Z-Score)
Description: Z-scores are calculated using Centers for Disease Control and Prevention (CDC) Growth Charts. Change from baseline was defined as the values for Z-score at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to study treatment administration. Negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | All Participants
Number analyzed (Participants) | 66
Z-score
  Month 6 | 0.0734 (0.1433)
  Month 12: number analyzed (Participants) | 65
  Month 12 | 0.0204 (0.1567)

8. Secondary Outcome: Change From Baseline in Percentile for Height for Age
Description: Z-scores were calculated using CDC growth charts, that contained Box-Cox transformation (L), the median (M) and the generalized coefficient of variation (S). Percentile was obtained using the following equation M (1 + LSZ) ** (1/L), where ** indicated an exponent, such that m (1+LSZ)** (1/L) meant raising (1+LSZ) to the (1/L)th power and then multiplying the M. Z was the Z-score that corresponds to the percentile. Negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline was defined as the values for percentile of Z-score at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentiles of Z-score
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentiles of Z-score
  Month 6 | 1.4675 (2.8638)
  Month 12 | 0.2810 (3.2237)

9. Secondary Outcome: Change From Baseline in Growth Velocity
Description: Growth velocity analysis was part of auxological parameter. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeter (cm)/year
Arm/Group | All Participants
Number analyzed (Participants) | 66
centimeter (cm)/year
  Month 6: number analyzed (Participants) | 65
  Month 6 | -3.938 (6.075)
  Month 12: number analyzed (Participants) | 63
  Month 12 | -4.798 (5.577)

10. Secondary Outcome: Percentage of Participants With Bone Age (BA)/Chronological Age (CA) Ratio Not Risen
Description: BA was determined using X-rays of the hand and wrist by Greulich and Pyle method. CA was calculated as (visit date -birth date + 1)/365.25. Percentage of response was calculated as n/N*100, where n was number of participants in the specified category and N was number of participants in the analysis population.
Time Frame: At Months 6 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentage of participants
  Month 6 | 95.5 [87.3 to 99.1]
  Month 12: number analyzed (Participants) | 65
  Month 12 | 92.4 [83.2 to 97.5]

11. Secondary Outcome: Change From Baseline in BA:CA Ratio
Description: BA was determined using X-rays of the hand and wrist by Greulich and Pyle method. CA was calculated as (visit date -birth date + 1)/365.25. Change from baseline was defined as the values for BA:CA ratio at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Participants
Number analyzed (Participants) | 66
ratio
  Month 6 | -0.04 (0.06)
  Month 12: number analyzed (Participants) | 65
  Month 12 | -0.06 (0.07)

12. Secondary Outcome: Percentage of Participants With Stabilized Pubertal Stage
Description: Pubertal stage parameters were analyzed using Tanner method. Pubertal stage parameters included genital development stage (GDS) in male participants, breast development stage (BDS) in female participants and pubic hair development (PHD) stage in both sexes. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Months 6 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
percentage of participants
  BDS for female participants, Month 6: number analyzed (Participants) | 62
  BDS for female participants, Month 6 | 98.4 [91.3 to 100.0]
  GDS for male participants, Month 6: number analyzed (Participants) | 4
  GDS for male participants, Month 6 | 100 [39.8 to 100.0]
  PHD for female participants, Month 6: number analyzed (Participants) | 62
  PHD for female participants, Month 6 | 91.9 [82.2 to 97.3]
  PHD for male participants, Month 6: number analyzed (Participants) | 4
  PHD for male participants, Month 6 | 100 [39.8 to 100.0]
  BDS for female participants, Month 12: number analyzed (Participants) | 61
  BDS for female participants, Month 12 | 93.5 [84.3 to 98.2]
  GDS for male participants, Month 12: number analyzed (Participants) | 4
  GDS for male participants, Month 12 | 100 [39.8 to 100.0]
  PHD for female participants, Month 12: number analyzed (Participants) | 61
  PHD for female participants, Month 12 | 87.1 [76.1 to 94.3]
  PHD for male participants, Month 12: number analyzed (Participants) | 4
  PHD for male participants, Month 12 | 75.0 [19.4 to 99.4]

13. Secondary Outcome: Percentage of Participants With Regression of Uterine Length
Description: Uterine length was determined by transabdominal ultrasound. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Months 6 and 12
Population: The ITT population consisted of all participants who received at least 1 dose of study intervention. Only data from the female participants analyzed were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
percentage of participants
  Month 6: number analyzed (Participants) | 57
  Month 6 | 64.5 [51.3 to 76.3]
  Month 12: number analyzed (Participants) | 54
  Month 12 | 64.5 [51.3 to 76.3]

14. Secondary Outcome: Percentage of Participants With Absence of Progression of Testis Volumes
Description: Testis volume was a clinical assessment with orchidometer. Percentage of response was calculated by number of participants in the specified category divided by number of participants in the analysis population multiplied by 100.
Time Frame: At Months 6 and 12
Population: The ITT population consisted of all participants who received at least 1 dose of study intervention. Only data from the male participants analyzed were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 4
percentage of participants
  Month 6 | 75.0 [19.4 to 99.4]
  Month 12 | 75.0 [19.4 to 99.4]

15. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: BMI analysis was part of auxological parameter assessment. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilogram (kg)/meter square
Arm/Group | All Participants
Number analyzed (Participants) | 66
kilogram (kg)/meter square
  Month 6 | 0.282 (0.882)
  Month 12: number analyzed (Participants) | 65
  Month 12 | 1.195 (1.196)

16. Secondary Outcome: Change From Baseline in Weight
Description: Weight analysis was part of auxological parameter assessment. Change from baseline was defined as the value for each auxological parameter at indicated timepoints minus the value at baseline. Baseline was defined as the last non-missing measurement taken prior to the first study treatment administered.
Time Frame: Baseline and at Months 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | All Participants
Number analyzed (Participants) | 66
kg
  Month 6 | 2.020 (1.927)
  Month 12: number analyzed (Participants) | 65
  Month 12 | 5.146 (2.816)

17. Secondary Outcome: Plasma Concentrations of Triptorelin
Description: Blood samples were collected at specified timepoints.
Time Frame: Day 1, 4 hours post-injection; Month 3; Month 6, predose; Month 6, 4 hours post-injection; and Month 12
Population: The Pharmacokinetic (PK) set consisted of all participants who received at 1 dose of study treatment and had at least 1 valid triptorelin concentration. Only data from the participants analyzed were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | All Participants
Number analyzed (Participants) | 66
ng/mL
  Day 1, 4 hours post-injection | 41.8 (56.9)
  Month 3: number analyzed (Participants) | 63
  Month 3 | 0.0434 (76.8)
  Month 6, predose: number analyzed (Participants) | 46
  Month 6, predose | 0.0251 (648.7)
  Month 6, 4 hours post-injection: number analyzed (Participants) | 61
  Month 6, 4 hours post-injection | 24.7 (66.0)
  Month 12: number analyzed (Participants) | 50
  Month 12 | 0.0223 (110.3)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from the first dose of study treatment (Day 1) up to a maximum of approximately 344 days.
Description: The Safety population consisted of all participants who received at least 1 dose of study treatment and have at least 1 post-baseline safety assessment.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 59/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=66)
Pyrexia (General disorders) | 9 (9)
Influenza like illness (General disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Nocturnal emission (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Listless (Psychiatric disorders) | 1 (1)
Weight increased (Investigations) | 9 (9)
Urinary occult blood positive (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Eosinophil count increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Myoglobin blood increased (Investigations) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Asthenopia (Eye disorders) | 2 (2)
Refraction disorder (Eye disorders) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Mouth ulceration (Gastrointestinal disorders) | 2 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 31 (45)
COVID-19 (Infections and infestations) | 10 (10)
Suspected COVID-19 (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4)
Tonsillitis (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 7 (7)
Obesity (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT05029622/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT05029622/SAP_001.pdf